CLINICAL TRIAL: NCT02870725
Title: A Cognitive Behavioral Therapy (CBT) Depression Intervention in Persons With Co-Occurring Chronic Headache
Brief Title: CBT Depression Intervention for Co-Occurring Chronic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Ashley J. Britton, Doctoral Candidate, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002322
Record Dates: First submitted 2016-02-02; First posted 2016-08-17 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Depression; Headaches Chronic; Migraine Disorders
Keywords: chronic headaches, migraines, depression
MeSH Terms: conditions — Depression; Headache Disorders; Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Treatment As Usual) (No Intervention): Individuals randomized into the control condition will not receive any active treatment but will have access to customary, community-based supportive services. These individuals will complete the pre-, post- and 4-week post-intervention outcome assessment measures and will serve as a means of comparison for those in the other arm of the study.
- CBT Individual Psychotherapy (Treatment) (Experimental): Behavioral Intervention (Individual Psychotherapy). These individuals will complete the pre-, post- and 4-week post-intervention outcome assessment measures and will serve as a means of determining whether or not the intervention was effective compared to the control arm.
  Interventions: Behavioral: CBT Individual Psychotherapy

INTERVENTIONS:
Behavioral: CBT Individual Psychotherapy — The 4-session CBT treatment will include receipt of a manualized cognitive behavioral intervention, delivered individually, to treat the depression symptoms (e.g. cognitive restructuring, behavioral activation) and teach adaptive coping strategies to manage their depression. Ideally, the intervention will also positively affect their chronic headaches (i.e. reduction of headache frequency, severity and level of disability). Each session is approximately 60 minutes with specific, reflective and guided activities related to a specific module within the intervention.
  Arms: CBT Individual Psychotherapy (Treatment)

SUMMARY:
Having co-occurring depression and chronic headaches is challenging and can greatly impact one's professional, personal, family, and social life. People living with chronic headaches are often at a greater risk of having comorbid psychiatric disorders (depression, anxiety), reduced quality of life, and impaired functioning because of under-diagnosis, misdiagnosis or under-treatment of both chronic conditions.

This study is a pilot clinical trial that will compare the effectiveness of a brief cognitive-behavior therapy (CBT) depression intervention to a care as usual (control) group. The aim of the study is to determine how well the CBT intervention will reduce the frequency, severity and level of disability of both the headaches and depression symptoms.

DETAILED DESCRIPTION:
STUDY LOCATIONS:

(A) University of Georgia College of Education in Athens, GA

(B) Henry Ford Hospital - Main campus in Detroit, MI.

* For the MI participants, you must be willing to travel to Detroit for the intervention if you choose to participate and are assigned to the treatment group.

**Please contact me with any questions about the study.**

Background: This research focuses on emphasizing alternative treatment approaches to underserved and marginalized groups. This study is a randomized pilot intervention to treat a community sample with co-occurring depression and chronic pain (i.e. headaches/migraines) - since they are at an increased risk for impaired functioning, comorbid psychiatric disorders and reduced quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age & living in GA or MI;
* a PHQ-9 score ≥5; AND
* have frequent migraines and/or moderate to severe headaches = 10 or more headache days per month for the past 3 months
* May or may not be taking headache/migraine medication so long as still meet other criteria
* ** For MI participants: must be willing & able to come to Detroit campus for the intervention (4 weeks in a row)

Exclusion Criteria:

* outside of 18-75 year old age range;
* Do not live in GA or MI
* Unable or unwilling to drive to campus location for the 4 sessions (treatment group only)
* do not have both conditions of depression and frequent/near-chronic headaches
* Active suicidal ideation (detailed plan and/or access to lethal means) or suicide attempts within the past 60 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Mean change in "Beck Depression Inventory (BDI-2)" | Initial 4-week change from pre-intervention to post-intervention & at 4-week post-intervention follow-up
  A 21-item likert scale developed to assess the intensity of depression while also monitoring changes over time.
Mean change in "Headache Disability Index" | Initial 4-week change from pre-intervention to post-intervention & at 4-week post-intervention follow-up
  A 27-item measure that assesses the impact of headache on daily living, headache treatment and the level of disability experienced.

SECONDARY OUTCOMES:
Mean change in "Migraine Disability Assessement Questionnaire (MIDAS)" | Initial 4-week change from pre-intervention to post-intervention & at 4-week post-intervention follow-up
  A 7-item questionnaire developed to assess the severity of disability related to migraines within the past 3 months, in 3 domains: school/paid work, household chores, & family/social/leisure activities
Mean change in "Headache Management Self-Efficacy Scale Adapted for Recurrent Headaches (HSES)" | Initial 4-week change from pre-intervention to post-intervention & at 4-week post-intervention follow-up
  A 25-item likert scale developed for recurrent headache sufferers to assess an individual's self-efficacy in preventing their headaches.
Mean change in "Headache Specific Locus of Control (HSLoC)" | Initial 4-week change from pre-intervention to post-intervention & at 4-week post-intervention follow-up
  A 33-item Likert scale designed to assess an individual's perceptions (locus of control) about their headache problems and headache relief on 3 dimensions: individual behavior (internal factor), healthcare professionals (external factor), or chance factors.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette D Heckman, PhD, Study Chair — University of Georiga; Benilda P Pooser, Study Director — University of Georgia, VP office for research
Locations (2):
- United States (2):
  - University of Georgia, Athens, Michigan
  - Henry Ford Hospital, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available. Only the dummy coded data set will be shared between UGA and HFHS for statistical analysis. Results will be discussed from an aggregate data perspective.

REFERENCES:
- [Background] Baskin SM, Lipchik GL, Smitherman TA. Mood and anxiety disorders in chronic headache. Headache. 2006 Oct;46 Suppl 3:S76-87. doi: 10.1111/j.1526-4610.2006.00559.x. PMID 17034402
- [Background] Weeks RE. Application of behavioral therapies in adult and adolescent patients with chronic migraine. Neurol Sci. 2013 May;34 Suppl 1:S11-7. doi: 10.1007/s10072-013-1360-6. PMID 23695037
- [Background] Martin P., Meadows G., Piterman L., Sharman M., Reece J., & Milgrom J. Cognitive Behavioral Therapy Effective for Comorbid Chronic Headache, Depression. Retrieved December 23, 2014, from http://www.psychcongress.com/article/cognitive-behavioral-therapy-effective-comorbid-chronic-headache-depression-12514, 2013.
- [Background] Nimnuan C., & Srikiatkhachorn A. Migraine: Psychiatric comorbidities. Retrieved January 25, 2015, from http://www.medmerits.com/index.php/article/migraine_psychiatric_comorbidities, 2011.
- [Background] Saper JR. Pearls from an inpatient headache unit. Headache. 2008 Jun;48(6):820-7. doi: 10.1111/j.1526-4610.2008.01141.x. PMID 18549359
- [Background] Shapiro R, Goadsby P. The long drought: the dearth of public funding for headache research. Cephalalgia. 2007 Sep;27(9):991-4. doi: 10.1111/j.1468-2982.2007.01396.x. No abstract available. PMID 17727471
- [Background] Muñoz, R. & Miranda, J. (1986, Revised 1993). Group Therapy Manual for Cognitive-behavioral Treatment of Depression. San Francisco General Hospital, Depression Clinic. Available from the author. University of California, San Francisco, Department of Psychiatry, San Francisco General Hospital, 1001 Potrero Avenue, Suite 7M, San Francisco, CA 94110.
- [Result] Breslau N, Lipton RB, Stewart WF, Schultz LR, Welch KM. Comorbidity of migraine and depression: investigating potential etiology and prognosis. Neurology. 2003 Apr 22;60(8):1308-12. doi: 10.1212/01.wnl.0000058907.41080.54. PMID 12707434
- [Result] Castien RF, van der Windt DA, Dekker J, Mutsaers B, Grooten A. Effectiveness of manual therapy compared to usual care by the general practitioner for chronic tension-type headache: design of a randomised clinical trial. BMC Musculoskelet Disord. 2009 Feb 12;10:21. doi: 10.1186/1471-2474-10-21. PMID 19216763
- [Result] Frediani F, Villani V. Migraine and depression. Neurol Sci. 2007 May;28 Suppl 2:S161-5. doi: 10.1007/s10072-007-0771-7. PMID 17508165
- [Result] Hamelsky SW, Lipton RB. Psychiatric comorbidity of migraine. Headache. 2006 Oct;46(9):1327-33. doi: 10.1111/j.1526-4610.2006.00576.x. PMID 17040330
- [Result] Sammons M. Treatment of head pain with psychotropics. Professional Psychology: Research and Practice, 36(6): 611-614, 2005.
- [Result] Shulman, R. (2013, May 17). Psychiatric Aspects of Headache, Pain and Depression [Webinar]. In National Headache Foundation Webinar Series. Retrieved January 30, 2015 from https://www.youtube.com/watch?v=4n3BTs6-fFU&list=PL6bpjkbYtk-MBnNjRF7pAxzBJI52_XdPd.
- [Result] Smitherman TA, McDermott MJ, Buchanan EM. Negative impact of episodic migraine on a university population: quality of life, functional impairment, and comorbid psychiatric symptoms. Headache. 2011 Apr;51(4):581-9. doi: 10.1111/j.1526-4610.2011.01857.x. PMID 21457242